CLINICAL TRIAL: NCT03926754
Title: Beta 3 Agonist Treatment in Heart Failure-2
Acronym: BEAT-HF II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Henning Bundgaard (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Hillerød hospital, Denmark (Unknown); Herlev Hospital (Other); Hvidovre University Hospital (Other); Bornholm Hospital, Denmark (Unknown); Royal North Shore Hospital (Other)
Responsible Party: Sponsor-Investigator, Henning Bundgaard, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-002367-34; H-16030780 (Other: Regional Ethics Committee)
Record Dates: First submitted 2017-07-04; First posted 2019-04-24 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction NYHA Class III-IV
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirabegron (Active Comparator): Active treatment arm (mirabegron)
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Study A The maximum tolerated dose up to a maximum of 300 mg per day for 26 weeks.
  Study B One single dose of 300 mg at day one followed by 150 mg x 2 for 1 week (8-11 days).
  Other Names: Placebo

SUMMARY:
Objective: The objective of the study is to assess the structural and functional cardiac effects of treatment with the beta 3 AR agonist Mirabegron in patients with moderate to severe chronic heart failure (LVEF<35%, NYHA III-IV).

The study is a randomized, placebo-controlled, double-blinded trial in two phases with two hypotheses:

Chronic study - study A: Long-term treatment (3 months) with the β3 adrenergic receptor agonist Mirabegron is beneficial in patients with moderate to severe human heart failure

Invasive study - Study B: Administration of Mirabegron in patients with heart failure leads to an immediate increase in cardiac output at a constant or reduced left ventricular filling pressure during submaximal exercise

Specific aims

1. Determine safety of administration of Mirabegron to patients with moderate to severe heart failure.
2. Determine if treatment with Mirabegron for 3 months induces beneficial cardiac structural remodelling in patients with moderate to severe heart failure. In an open-label follow-up to determine the effects of Mirabegron after an extended duration (a total of 12 months).
3. Determine if Mirabegron improves symptoms and exercise capacity as indicated by questionnaires and 6 min walk test in patients with moderate to severe heart failure.
4. Determine effects of Mirabegron on cardiac conduction, repolarisation and rhythms and arrhythmias in patients with moderate to severe heart failure.
5. Determine effects of Mirabegron on circulating biomarkers in patients with moderate to severe heart failure.
6. Determine the immediate and short term haemodynamic effects of Mirabron as measured by CT and invasively.

ELIGIBILITY:
Inclusion Criteria:

1. Stable heart failure NYHA class III-IV on ischemic or non-ischemic basis
2. Left ventricular ejection fraction (LVEF) < 35% as assessed by cardiac CT
3. NT proBNP > 1000 pg/ml
4. On optimised evidence-based pharmacological HF treatment stable ≥2 weeks with no current plan for changing HF therapy. The therapy must include a beta-blocker.
5. No change in diuretics ≤1 week
6. No admittances to hospital for treatment with intravenously administered positive inotropic agents ≤ 4 weeks.
7. >18 years

Exclusion Criteria:

1. Acute myocardial infarction (AMI) or revascularisation < 3 month ago
2. Uncorrected significant primary obstructive valve disease
3. Planned major surgery including cardiac revascularisation
4. Hemodynamically significant obstructive cardiomyopathy
5. Acute myocarditis or constrictive pericarditis
6. Clinically significant hepatic (transaminases or bilirubin x 3 above upper reference level) or renal (GFR< 30 ml/min/1,73 m2) diseases
7. Heart failure due to uncorrected thyroid disease
8. Cardiac mechanical support
9. < 6 months after CRT
10. Uncontrolled hypotension (defined as symptomatic systolic blood pressure < 80 mmHg) - or hypertension (defined as systolic at 180 mmHg or above and/or diastolic blood pressure at 110 mmHg or below)
11. Unable to give informed consent
12. Reduced compliance
13. All women of child bearing potential will be required to use adequate contraception
14. Pregnant or lactating women
15. Treatment with a tricyclic antidepressant or CYP2D6 substrates other than beta-blockers or treatment with digoxin.
16. Known allergy to iodine containing contrast
17. Estimated GFR < 30 ml/min/1.73 m2
18. Congenital or drug induced QT prolongation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Increase in left ventricular ejection fraction as measured by computed tomography | 3 months
  Study A
Change in invasive hemodynamics assesses by right heart catherization | At 3 hours and at 1 week
  Study B is explorative assessing the effect on invasive parameters including cardiac output, pulmonary wedge pressure and pulmonary and systemic vascular resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Because of the sensitive nature of the data collected for this study, requests to access the dataset from qualified researchers trained in human subject confidentiality protocols may be sent to the principal investigator.

REFERENCES:
- [Background] Bundgaard H, Axelsson A, Hartvig Thomsen J, Sorgaard M, Kofoed KF, Hasselbalch R, Fry NA, Valeur N, Boesgaard S, Gustafsson F, Kober L, Iversen K, Rasmussen HH. The first-in-man randomized trial of a beta3 adrenoceptor agonist in chronic heart failure: the BEAT-HF trial. Eur J Heart Fail. 2017 Apr;19(4):566-575. doi: 10.1002/ejhf.714. Epub 2016 Dec 18. PMID 27990717